CLINICAL TRIAL: NCT05000983
Title: A Between Patient, Pilot Randomized Controlled Study of Plurogel® Compared to Standard Topical Dressing in Burn Injuries
Brief Title: A Between Patient Study of Plurogel® Compared to Standard Topical Dressing in Burn Injuries
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: between
Record Dates: First submitted 2021-05-19; First posted 2021-08-11 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Burns
Keywords: burn; wound; debridement
MeSH Terms: conditions — Burns; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard dressing (Active Comparator): Topical antibiotic ointment (Polysporin™ or formulary equivalent) and non-adherent petrolatum fine-meshed gauze (ADAPTIC™) applied every Monday, Wednesday and Friday (or equivalent).
  Interventions: Drug: Standard dressing
- Test dressing (Experimental): A 0.5 cm layer of PluroGel® followed by the above standard dressing. In addition, this will be covered with moistened gauze, kept moist twice daily. (The additional factors are the use of PluroGel® and moistened gauze. Standard dressing will continue to be used.)
  Interventions: Drug: PluroGel

INTERVENTIONS:
Drug: PluroGel — A 0.5 cm layer of PluroGel® followed by the above standard dressing. In addition, this will be covered with moistened gauze, kept moist twice daily. (The additional factors are the use of PluroGel® and moistened gauze. Standard dressing will continue to be used.)
  Arms: Test dressing
Drug: Standard dressing — Topical antibiotic ointment (Polysporin™ or formulary equivalent) and non-adherent petrolatum fine-meshed gauze (ADAPTIC™) applied every Monday, Wednesday and Friday (or equivalent).
  Arms: Standard dressing

SUMMARY:
Burn injuries can result in long term physical and mental sequelae, not only from the scarring but also the painful dressings. The standard of care today remains use of antibiotic topical dressings while awaiting demarcation of the burn depth, with surgical excision and grafting for deep partial thickness and full thickness areas. Demarcation can be appreciated on admission for full thickness burns but is often a prolonged process that can last weeks. The clinical evaluation of the depth of the burn is a complex decision that often is made more challenging by the presence of the proteinaceous pseudoeschar and the coagulated dermis itself. Surgical debridement is relatively 'coarse' and by its very nature requires removal of a thin layer of viable tissue to reach the level that is vascularized enough to support a skin graft. There has been growing interest in the use of adjuncts to reduce the amount tissue debrided and potentially reduce the need for surgery itself. Operatively, there have been some reports that use of hydro-dissection devices (Versajet™) may allow a more controlled debridement, resulting in less viable tissue being sacrificed. There is also a growing experience with enzymatic debridement, especially with Bromolein, derived from Pineapple (NexoBrid®). Neither of these have been shown to definitively improve care in randomized controlled trials, (RCTs) and there is suggestion that in some settings may actually cause harm.

DETAILED DESCRIPTION:
Burn injuries can result in long term physical and mental sequelae, not only from the scarring but also the painful dressings. The standard of care today remains use of antibiotic topical dressings while awaiting demarcation of the burn depth, with surgical excision and grafting for deep partial thickness and full thickness areas. Demarcation can be appreciated on admission for full thickness burns but is often a prolonged process that can last weeks. The clinical evaluation of the depth of the burn is a complex decision that often is made more challenging by the presence of the proteinaceous pseudoeschar and the coagulated dermis itself. Surgical debridement is relatively 'coarse' and by its very nature requires removal of a thin layer of viable tissue to reach the level that is vascularized enough to support a skin graft. There has been growing interest in the use of adjuncts to reduce the amount tissue debrided and potentially reduce the need for surgery itself. Operatively, there have been some reports that use of hydro-dissection devices (Versajet™) may allow a more controlled debridement, resulting in less viable tissue being sacrificed. There is also a growing experience with enzymatic debridement, especially with Bromolein, derived from Pineapple (NexoBrid®). Neither of these have been shown to definitively improve care in randomized controlled trials, (RCTs) and there is suggestion that in some settings may actually cause harm.

A relatively recent entry into the 'space' of non-surgical burn wound debridement is Plurogel®. Unlike Bromolein, Plurogel® is a concentrated surfactant in the form of a stable, viscous gel. Each micelle has a hydrophilic outer surface that softens and loosens wound debris, and a hydrophobic inner core that traps debris. The micelles link to form a matrix that continually expands and contracts. This creates a cleansing/rinsing action that disrupts the surface tension holding slough and necrotic tissue in place. PluroGel® helps in creating a moist wound healing environment, which softens, loosens and drives slough and necrotic debris away from the wound bed, promoting autolytic debridement. PluroGel® is approved for use in burn injuries in Canada, however there are no randomized control trials (RCTs) to support its use. As Plurogel® appears to fill a much-needed niche in burn wound care, and as our centre seeks to be innovative in patient care, we trialed Plurogel® on some of our appropriately consented burn patients. The anecdotal experience is that the eschar lifted within about a week and there was visible wound healing. Healing time appeared to be reduced as the product would gently debride while still providing a moist wound bed encouraging wound healing. Team members began to value the new product. This early positive experience is the impetus for us to embark on a pilot RCT to provide evidence for us to continue to use this product.

ELIGIBILITY:
Inclusion Criteria:

* Persons with partial thickness face burns or unilateral limb burn injuries requiring admission.

Exclusion Criteria:

* Total burn surface area (TBSA) >30%.
* Burn depth full thickness or deeper on initial assessment.
* Prior excision at another healthcare centre.
* Patients with pre-existing malnutrition
* Electrical, chemical or other unusual burn etiologies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | 1-14 days
  Days to over 80% area of burn injury healed

SECONDARY OUTCOMES:
Patient and caregiver satisfaction and perception of pain | At each dressing change
  Measure satisfaction and perception of pain using a survey
Proportion requiring surgery | 1-14 days
  Proportion of burn injuries that require skin grafting in each group
Relative surface area skin grafted | 1-14 days
  Calculate area of burn needing grafting and area of burn that does not need graft

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No